CLINICAL TRIAL: NCT05291416
Title: Sarcopenia; a New Issue in Juvenile Idiopathic Arthritis
Brief Title: Sarcopenia in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, lassoued ferjani Hanene, Assistant professor, University Tunis El Manar
Other Study IDs: pediatric rheumatology Kassab
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia; Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Sarcopenia; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: healthy children aged between 4-16 years
  Interventions: Diagnostic Test: densitometry/ handgrip dynamometer
- 2: children aged between 4-16 years, suffering from juvenile idiopathic arthritis
  Interventions: Diagnostic Test: densitometry/ handgrip dynamometer

INTERVENTIONS:
Diagnostic Test: densitometry/ handgrip dynamometer — all patients will undergo the Dual-energy X-ray absorptiometry (DXA) and the muscle strength assessment using the handgrip dynamometer

SUMMARY:
Juvenile idiopathic arthritis (AJI), is a frequent inflammatory disease in children, characterized by pain, arthritis, and deformities. Chronic inflammation leads to physical inactivity and can be associated with muscle weakness around affected joints, low bone strength, and mass(3). To our knowledge, no study has focused on the prevalence of sarcopenia in JIA and the data on the muscle disorder are lacking. The purpose of the present study is to detect sarcopenia and identify associated factors in children with JIA

ELIGIBILITY:
Inclusion Criteria:

* children with juvenile idiopathic arthritis fulfilling the ILAR criteria

Exclusion Criteria:

* We excluded patients who have a prosthesis, nutritional problems, inflammatory bowel disease, coeliac disease, temporomandibular involvement, or another chronic disease.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For all patients, we collected the anthropometric data including weight, height, and expressed it as Z scores for age and sex. Body mass index (BMI) was calculated as weight (kg)/height (m2). The disease duration, AJI subtype, disease activity, and treatment were recorded.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
skeletal muscle mass | 4 months
  Dual-energy X-ray absorptiometry (DXA) measures the appendicular lean mass ( the sum of the lean mass of the arms and legs) and adjusted to the body mass index

SECONDARY OUTCOMES:
muscle strenght | 5 months
  Three consecutive trials will be measured by the handgrip dynamometer between the dominant and non-dominant sides. the highest value will be used and adjusted to the body mass index

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lassoued Ferjani H, Majdoub F, Ben Nessib D, Kaffel D, Triki W, Maatallah K, Hamdi W. Sarcopenia: a new issue in juvenile idiopathic arthritis. A study Protocol. Tunis Med. 2023 Jan 2;101(1):15-18. PMID 37682255